CLINICAL TRIAL: NCT03511677
Title: Effectiveness of Insole on Morton's Neuroma
Brief Title: Insole on Morton's Neuroma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Hilda Alcantara Veiga de Oliveira, PT, MsC, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20634013.9.0000.5505.
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Morton Neuroma
Keywords: Insole; Morton Neuroma; Pain; Function
MeSH Terms: conditions — Morton Neuroma; Pain | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo insole
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Customized insole with metatarsal support
  Interventions: Device: Insole
- Control Group (Placebo Comparator): Placebo flat insole
  Interventions: Device: Placebo Insole

INTERVENTIONS:
Device: Insole — Customized insole
  Arms: Intervention Group
Device: Placebo Insole — Placebo flat insole
  Arms: Control Group

SUMMARY:
Objective: The aim of the present study was to assess the effectiveness of insole with metatarsal support on pain in patients with Morton's neuroma and the impact of this insole on function, load distribution in the plantar region, gait variables, quality of life and satisfaction with insole use.

Methods: A randomized, controlled, double-blind, clinical trial with intent-to-treat analysis. Seventy-two patients with Morton's neuroma were randomly allocated into a study group and control group. One week following the baseline evaluation, the study group received insole with metatarsal support made of ethyl vinyl acetate and the control group received a flat insole of the same material, color and density. The groups were evaluated after 6, 12 and 24 weeks of insole use. The following assessment parameters employed: pain when walking and at rest (END); quality of life (SF-36); foot function (FFI and FHSQ); six-minute walk test (6MWT) and foot pressure analysis using the AM Cube FootWalk Pro program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical and radiological diagnosis (magnetic resonance or ultrasound) of Morton's neuroma.
* Pain in the foot with VAS between 3-8 cm to walk.
* Over 18 years.
* No distinction of sex
* Agree to participate of the study and sign the informed consent form.

Exclusion Criteria:

* Other symptomatic musculoskeletal diseases in MMII.
* Symptomatic diseases of the central and peripheral nervous system.
* Diabetes Mellitus.
* Rigid deformities on foot.
* Use of insoles in the last three months.
* Physiotherapy in the last three months.
* Infiltrations on foot and ankles in the last three months.
* Previous or expected surgery in the next twelve months.
* Allergy to the material of the insole.
* Mental deficiency.
* Geographic inaccessibility .- Use of corticosteroids or NSAIDs in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline, after 6, 12 and 24 weeks
  Measured by visual analogue scale from 0 cm to 10 cm

SECONDARY OUTCOMES:
Change in function and foot health | Baseline, after 6, 12 and 24 weeks
  Measured by Foot function index questionnaire
Change in function, foot healt and quality of life | Baseline, after 6, 12 and 24 weeks
  Measured by Foot Health Status questionnaire
Change in function | Baseline, after 6, 12 and 24 weeks
  Measured by the distance in the six minute walking test
Quality of life | Baseline, after 6, 12 and 24 weeks
  Measured by the Short Form -36 questionnaire

IPD SHARING:
Plan to Share IPD: No